CLINICAL TRIAL: NCT00692484
Title: Pilot Evaluation of the Effect of Application Procedure on the Antimicrobial Effects of an Aqueous CHG and a Traditional Iodophor Scrub Paint
Brief Title: Pilot Evaluation of the Application Procedure on the Antimicrobial Effects of 2 Antiseptics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 060629
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Healthy
Keywords: Antimicrobial; Antisepsis; Topical antisepsis
MeSH Terms: interventions — chlorhexidine gluconate; Povidone-Iodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Chlorhexidine gluconate 2%
  Interventions: Drug: Chlorhexidine gluconate
- 2 (Active Comparator): Povidone iodine scrub and paint
  Interventions: Drug: Povidone iodine

INTERVENTIONS:
Drug: Chlorhexidine gluconate — Chlorhexidine gluconate (2% w/v) in an aqueous base. Administered topically.
  Other Names: ChloraPrep AQ
  Arms: 1
Drug: Povidone iodine — Povidone iodine scrub and paint. Administer topically.
  Other Names: Betadine
  Arms: 2

SUMMARY:
Evaluate effect of application procedure on efficacy of 2 antiseptics for cleaning skin prior to surgery.

DETAILED DESCRIPTION:
Evaluate the effect of application procedure on the antimicrobial properties of a new product and a currently marketed product. Study will be conducted using methods dictated by the FDA.

Study uses topical sampling from the abdomen and groin on intact skin and evaluates the germs. Effects of blotting versus not blotting will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Free of dermatoses, cuts, lesions, or other skin disorders around test sites
* must not have received topical or systemic antimicrobials, antibiotics, or steroids for 7 days prior to testing and agree to abstain from these materials until completion of the study

Exclusion Criteria:

* Exposure of test sites to antimicrobial agents, medicated soaps, medicated shampoos, or medicated lotions, use of biocide-treated pools or hot tubs, use of tanning beds, or sunbathing during the 7 day pre-test period or during the test period
* exposure of the test sites to strong detergents, solvents, or other irritants during the 7 day pre-test period or during the test period
* use of systemic or topical antibiotic medications, steroid medications, or any other product known to affect the normal microbial flora of the skin during the 7 day pre-test period or during the test period
* known allergy to latex (rubber), alcohols, inks, or tape adhesives, or to common antibacterial agents found in soaps, lotions, or ointments, particularly chlorhexidine gluconate and povidone iodine
* active skin rashes or breaks in the skin of the test sites
* currently active skin disease or inflammatory skin condition, including contact dermatitis
* showering or bathing within the 72 hour period prior to sampling
* participation in a clinical study in the past 7 days or current participation in another clinical study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2007-10; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
3.0 log10 reduction in CFU/cm2 on inguinal sites, and 2.0 log10 reduction in CFU/cm2 on abdominal sites | 10 minutes and 6 hours after application of test solutions

SECONDARY OUTCOMES:
Impact of blotting versus not blotting | Blotting and not blotting after 2 minute application with CHG and 5 minute application of iodophor

CONTACTS AND LOCATIONS:
Overall Officials: Daryl S Paulsen, PhD, Principal Investigator — President and CEO
Locations (1):
- BioScience Laboratories, Bozeman, Montana, United States